CLINICAL TRIAL: NCT03870620
Title: Metastatic Breast Cancer in Austria
Status: Recruiting | Type: Observational
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Hoffmann-La Roche (Industry); Daiichi Sankyo (Industry); Pfizer (Industry); Novartis (Industry); Caris Life Sciences (Industry); AstraZeneca (Industry); Seagen Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: AGMT_MBC-Registry
Record Dates: First submitted 2019-01-08; First posted 2019-03-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Breast Carcinoma; Breast Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Breast cancer is the most common cancer among women worldwide. In Austria, this diagnosis is made more than 5000 times a year (STATISTICS AUSTRIA, Austrian Cancer Registry, as of 24.09.2012). Of these, already 5% to 10% have distant metastases at the time of initial diagnosis, and up to 30% of the node-negative tumours and up to 70% of the node-positive tumours metastasise at a later date. Metastatic breast cancer has not been systematically assessed in Austria to date. This medical registry of the AGMT is thus the first Austrian-wide standardised documentation of this disease. The aim of the registry is to answer both epidemiological and therapy-specific questions.

This registry is a prospective and retrospective, multicentre collection of data on patients with metastatic breast cancer in Austria. All tumour characteristics, medical histories and also treatment sequences are documented in anonymised form.

DETAILED DESCRIPTION:
The present AGMT registry will provide accurate documentation of initial disease progression and initial tumour characteristics in patients with metastatic breast cancer in Austria. The data collected will include: median age at metastasis, median disease-free survival (DFS) between initial diagnosis or first date of absence of disease and occurrence of metastasis, histological subtype of the primary tumour, initial TNM stage, grade and receptor status of the primary tumour, type and form of adjuvant therapy, pattern of metastasis and metastasis site. Characteristics that have a negative prognostic value are expected to be overrepresented in the metastatic patient group.

Also, this AGMT registry is intended to assess the distribution pattern of these metastatic stage subtypes in Austria. Additionally, their influence on treatment strategy and outcome is to be studied. Furthermore, the frequency and tumour characteristics of breast cancer in male patients will be assessed and the influence of gender on treatment strategies identified.

The AGMT breast cancer registry will conduct an exact analysis of survival data, thereby enabling accurate calculations of average survival duration in patients with metastatic breast cancer in Austria. Further parameters that reflect the quality or course of oncological treatment are the survival rates from the time of metastasis development at 1, 2 and 5 years after diagnosis.

This AGMT registry is intended to investigate the response to various therapies in a real life population in relation to previous treatments, concomitant diseases and breast cancer subtype. The aim is to assess which therapies are used at which time point and on which disease subtype they depend.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of breast cancer
* Histological and/or radiological evidence of metastases
* Metastasis within 10 years of registry initiation
* Signed informed consent (if a patient has already died at the time of entry, the entry can be made without a declaration of consent)

Exclusion Criteria:

* Due to the non-interventional design of the registry there are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry is a prospective and retrospective, multicentre collection of data on patients with metastatic breast cancer in Austria.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-06-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with prognostic factors for metastatic breast cancer | 10 years
Number of patients according to molecular subtypes | 10 years
Frequency and tumour characteristics of breast cancer in male patients | 10 years
Overall survival of patients with metastatic breast cancer in Austria | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Study Chair — AGMT gemeinnützige GmbH
Locations (16):
- Austria (16):
  - Landeskrankenhaus Salzburg Universitätsklinikum der Paracelsus Medizinischen Privatuniversität; Universitätsklinik für Innere Medizin III Salzburg, Salzburg, Salzburg
  - Steiermärkische Krankenanstalten- gesellschaft m. b. H. LKH-Univ. Klinikum Graz; Universitätsklinik für Innere Medizin; Klinische Abteilung für Onkologie, Graz, Styria
  - Landeskrankenhaus - Universitätskliniken Innsbruck; Universitätsklinik für Frauenheilkunde Innsbruck, Innsbruck, Tyrol
  - BKH Kufstein; Innere Medizin: Interne II und onk. Tagesklinik, Kufstein, Tyrol
  - Kepler Universitätsklinikum; Univ.-Klinik für Hämatologie und Internistische Onkologie, Linz, Upper Austria
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern; Interne I: Medizinische Onkologie und Hämatologie, Linz, Upper Austria
  - Pyhrn-Eisenwurzen Klinikum Steyr; Innere Medizin II: Onkologie, Gastroenterologie, Angiologie, Steyr, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH; Abteilung für Innere Medizin IV, Wels, Upper Austria
  - AKH Wien; Universitätsklinik für Frauenheilkunde: Klin. Abt. f. Allg. Gynäkologie und gynäkologische Onkologie, Vienna, Vienna
  - LKH Feldkirch; Innere Medizin II/ Interne E (Hämatologie und Onkologie), Feldkirch, Vorarlberg
  - Krankenhaus St. Josef Braunau; Inneren Medizin 2, Braunau am Inn
  - Krankenhaus der Stadt Dornbirn; Brustgesundheitszentrum Dornbirn, Dornbirn
  - Steiermärkische Krankenanstalten- gesellschaft m.b.H. LKH Hochsteiermark; Department für Hämato-Onkologie, Leoben
  - Universitätsklinikum St. Pölten; Abteilung für Innere Medizin 1, Sankt Pölten
  - UK AKH Wien: Universitätsklinik für Innere Medizin I: Klinische Abteilung für Onkologie, Vienna
  - Klinik Ottakring; 1. Med. Abteilung, Zentrum f. Onkologie, Hämatologie und Palliativmedizin, Vienna